CLINICAL TRIAL: NCT02845284
Title: Enhanced HIV/Sexually Transmitted Infections and Pregnancy Prevention Study to Improve Adolescent Reproductive Health Services in Uganda
Brief Title: 'HI-4-TU' Study: Health Improvement for Teen Ugandans Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: MU-JHU CARE (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00061475
Record Dates: First submitted 2016-07-20; First posted 2016-07-27 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Pregnancy; Human Immunodeficiency Virus; Sexually Transmitted Diseases
Keywords: adolescent; reproductive health
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Routine Care (No Intervention): Group education/counseling from Antenatal clinic midwives, routine PMTCT, HIV C&T and family planning C&T services on request.
- Routine Care plus group support (Experimental): Routine Care plus enhanced group support
  Interventions: Behavioral: enhanced group support
- Routine Care plus individual support (Experimental): Routine Care plus enhanced individual support
  Interventions: Behavioral: enhanced individual support

INTERVENTIONS:
Behavioral: enhanced group support — Routine Care plus enhanced group support, and peer education beginning every 4 weeks post enrollment to delivery and at 6 and 10 weeks, 3, 6 and 9 months post delivery.
  Arms: Routine Care plus group support
Behavioral: enhanced individual support — Routine Care plus individual peer education and support beginning every 4 weeks post enrollment to delivery and at 6 and 10 weeks, 3, 6 and 9 months post delivery.
  Arms: Routine Care plus individual support

SUMMARY:
This randomized clinical trial is an adolescent focused implementation science study directed at improved social support and prevention of both HIV/STI's and subsequent unplanned pregnancies. The study population is pregnant adolescents who are attending antenatal care in Kampala, Uganda The acceptability and effectiveness of two enhanced peer lead, reproductive health promotion interventions compared to routine health care will be studied. The study participants will be individually randomized to one of three arms.

DETAILED DESCRIPTION:
The overall goal of this research to test the acceptability and effectiveness of two enhanced adolescent friendly reproductive health prevention interventions versus current routine care. In each intervention group, 152 adolescent mothers will be randomized to either the enhanced group peer support education and counseling intervention or to the enhanced one-to-one (individual) peer support education and counseling group with a young, model, peer educator trained to deliver Reproductive Health Education and counseling messages, beginning during pregnancy (≥ 28 weeks) and followed up to 9 months postpartum or study end at or after 6 months (whichever comes first). The control group will consist of 215 adolescent mothers randomized to routine care as provided at Mulago hospital (or the designated health facility) where midwives deliver group sessions during antenatal and postpartum care visits as well as standard PMTCT services including routine opt-out HIV C&T and availability of partner C&T. Syphilis testing should also be routinely provided and treatment provided for infected pregnant mothers and their partners as per local standard of care.

The 3 groups will be enrolled with study visits at 3, 6 and 9 months post partum however the intervention groups (Arms 2 and 3) will have additional visits at 36 weeks Antepartum, delivery, 6 and 10 weeks postpartum, Quantitative baseline data will be collected on routine demographic characteristics, reproductive history, pregnancy intentions and sexual risk/perceptions and HIV/Sexually Transmitted Infection status.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant at ≥28 weeks of gestation
* Agreeing to provide written informed consent to be screened for and take part in the study
* Agreeing to provide adequate locator information with residence within 30 km
* Agreeing to a home visit
* Agreeing to come for follow up visits and to receive study follow up phone calls

Exclusion Criteria:

* Serious illness or social conditions that would prevent adherence to study requirements
* High risk pregnancy or fetal death in utero (with the exception of risk defined only by maternal age)

Ages: 15 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 486 (Actual)
Dates: Start 2016-03-30 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Composite measure of consistent condom-use and use of an effective family planning method method | A comparison of this binary outcome will be conducted at one year.
  A log-binomial regression model will be used to obtain the prevalence rate ratios.
Incidence of any Sexually Transmitted Infection | at one year
  Kaplan-Meier survival analysis will be conducted to determine differences in the probability of sexually transmitted infection between study arms.

CONTACTS AND LOCATIONS:
Overall Officials: Florence Mirembe, MMED, PhD, Principal Investigator — MU-JHU Care Ltd
Locations (1):
- MUJHU CARE Ltd, Kampala, Wakiso DIstrict, Uganda

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT02845284/Prot_SAP_000.pdf